CLINICAL TRIAL: NCT01557374
Title: Tapering Abatacept or Tocilizumab in Rheumatoid Arthritis in Remission. An Evaluation of Disease Activity, Relapse Risk, Structural Progression and the Economic Impact of a Tapering Strategy
Brief Title: TOward the Lowest Effective DOse of Abatacept or Tocilizumab
Acronym: TOLEDO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AOM 11061
Record Dates: First submitted 2012-03-16; First posted 2012-03-19 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2020-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Disease activity; Remission; Lowest Effective DOse; Abatacept Tocilizumab; ACR-EULAR 2010
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Abatacept; Injections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Maintenance Tocilizumab, Abatacept (Active Comparator): No modification in biotherapy dose and administration frequency
  Interventions: Drug: Tocilizumab, Abatacept
- Decrease Tocilizumab, Abatacept (Experimental): Progressive decrease by predetermined pattern. Progressive injection interval increase (by stage)
  Interventions: Drug: Decrease Tocilizumab, Abatacept

INTERVENTIONS:
Drug: Tocilizumab, Abatacept — Tocilizumab: Roactemra 4-8 mg/kg/month and 162 mg/week Abatacept: Orencia 500-1000 mg/month and 125 mg/week
  Other Names: Tocilizumab: Roactemra 4-8 mg/kg/month (IV injections) and 162 mg/week (SC injections); Abatacept: Orencia 500-1000 mg/month (IV injections) and 125 mg/week (SC injections)
  Arms: Maintenance Tocilizumab, Abatacept
Drug: Decrease Tocilizumab, Abatacept — The decrease pattern is established on 4 consecutive stages :
  IV Abatacept (500-1000 mg/month) and Tocilizumab(4-8 mg/kg/month):
  Stage 0 : Perfusion /30 days Stage 1 :Perfusion/45 days Stage 2 :Perfusion/60 days Stage 3 :Perfusion/90 days Stage 4 :Stop
  SC Abatacept (125 mg/week) and Tocilizumab (162 mg/week):
  Stage 0 :Injection/7 days Stage 1 :Injection/10 days Stage 2 :Injection/14 days Stage 3 :Injection/21 days Stage 4 :Stop
  * If DAS 28 ≤ 2,6 (remission DAS persistent) on trimestrial visit: transfer to next stage for 3 months before next evaluation.
  * If DAS 28 > 2,6 et ≤ 3,2 (weak activity) : maintain ongoing stage
  * If DAS 28 > 3,2 : return to previous stage, (relapse according to European expert consensus)
  In the case of relapse while the patient is in stage 0, the therapy modification is left to the investigator's free will, but the patient will be followed till the end of the study.
  Other Names: Tocilizumab: Roactemra; Abatacept: Orencia
  Arms: Decrease Tocilizumab, Abatacept

SUMMARY:
Ever since the biotherapy agents have entered the market, the recommended therapeutic objective in Rheumatoid arthritis, has been remission. Once obtained, it is advised to try to reduce or cease these biotherapy agents, for which, their efficacy is counterbalanced to their tolerance in the medium and long term as well as their high price. Nevertheless, we do not dispose considerable data on the risks of relapse or structural progression during such a step down strategy. A few studies on anti-TNF agents have shown the possibility of such therapy reduction. A national study, " STRASS ", coordinated by Bruno FAUTREL, has evaluated the possibility of spacing or even stopping the injections of anti-TNF(s). To date, no data concerning Abatacept or Tocilizumab has been published.

As the expected result, this study is aimed to test the feasibility of a step down strategy on 2 biological agents, Abatacept and Tocilizumab, in RA patients in remission.

DETAILED DESCRIPTION:
Ever since the biotherapy agents have entered the market, the recommended therapeutic objective in Rheumatoid arthritis, has been remission. Once obtained, it is advised to try to reduce or cease these biotherapy agents, for which, their efficacy is counterbalanced to their tolerance in the medium and long term as well as their high price.

Nevertheless, we do not dispose considerable data on the risks of relapse or structural progression during such a step down strategy. A few studies on anti-TNF agents have shown the possibility of such therapy reduction. A national study, " STRASS ", coordinated by Bruno FAUTREL, has evaluated the possibility of spacing then stopping the injections of anti-TNF(s). To date, no data concerning Abatacept or Tocilizumab has been published.

This is a Non inferiority, prospective, randomized, controlled study with PROBE (Prospective Randomized, Open Blinded Evaluation) evaluating method.

The objectives of this study are:

* For patients with Rheumatoid Arthritis (RA) in remission under Abatacept or Tocilizumab, to evaluate in terms of disease activity within a 2 years period, the impact of a progressive decreasing biotherapy strategy (by progressively spacing the injections) in comparison with usual treatment (maintaining the usual dose and injection frequency of the biotherapeutic agent).
* To evaluate the impact of such decreasing strategy in terms of RA relapses and structural progression in 1 and 2 years.
* To determine the cost-effectiveness ratio of decreasing in comparison with maintaining the biological treatments.

Inclusion criteria:

Patients with RA, defined by ACR-EULAR 2010 criteria:

* Treated for at least 1 year with Abatacept or Tocilizumab with market authorized doses*, and possibly with a DMARD and ≤ 5 mg per day of corticoids.
* In remission for at least 6 months according to ACR/ EULAR 2010 remission criteria or a DAS 28 ≤ 2.6**

Patients are divided into 2 groups:

1. Maintaining strategy: to maintain the biological treatment and possibly the associated DMARD and corticoids.
2. Decreasing strategy: to decrease progressively the biological agent via progressively increasing the injection intervals, following a predetermined pattern, established according to the RA activity level, during each trimestrial visit.

The primary judgment criterion is: RA activity in a 2 years period of time, measured by repeated DAS44.

The secondary judgment criteria are:

* Percentage of relapse in 1 and 2 years.
* Radiographic structural progression in 1 and 2 years.
* Cost-effectiveness ratio difference between the 2 strategies in 2 years.

As the expected result, this study is aimed to test the feasibility of a step down strategy on 2 biological agents, Abatacept and Tocilizumab, in RA patients in remission.

ELIGIBILITY:
Inclusion Criteria:

* Patients of at least 18 years old.
* Patients with RA, defined by ACR-EULAR 2010 criteria
* Treated for at least 1 year with Abatacept or Tocilizumab with market authorized doses*, and possibly with a DMARD and ≤ 5 mg per day of corticoids.
* In remission since at least 6 months according to ACR/ EULAR 2010 remission criteria or a DAS 28 ≤ 2.6**
* Without destructive structural progression during the previous year on the hand and feet x-rays (judged by the reference rheumatologist)
* Informed on the study and have given their acknowledged written consent to participate in the study.
* Having had a prior medical visit.

  * Prescribed dose stability (a spacing related to an infection or a surgery is not a prescribed dose spacing).

    * An increase in inflammatory parameters and pain due to an intercurrent event must be distinguished from the RA activity increasing.

Exclusion Criteria:

* Already included in another treatment evaluation trial for the same pathology.
* Surgical intervention programmed for in the next 24 months to come.
* Pregnancy or it's anticipation in the next 24 months to come.
* Non comprehension of French language.
* Non affiliation to social security.
* Patients under legal guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
RA activity in a 2 years period of time, measured by repeated DAS44 | Trimestrial visit (-5 days/ + 35 days)
  The primary judgment criterion is: RA activity in a 2 years period of time, measured by repeated DAS44.

SECONDARY OUTCOMES:
Radiographic structural progression evaluation and cost-efficiency measure | 2 years
  RA relapse percentage in 1 and 2 years. Radiographic structural progression evaluation by annual radiography.(Sharp score) Cost- efficiency ratio difference between the 2 strategies of maintenance and decrease.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno FAUTREL, Pr, Principal Investigator — APHP
Locations (1):
- CHU Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided